CLINICAL TRIAL: NCT01475266
Title: Randomized, Placebo-controlled, Double-blinded Study of Single Immediate Instillation of EO9 After TURBT in Patients With NMIBC
Brief Title: Single Immediate Instillation of EO9 After TURBT in Patients With Non-muscle-invasive Bladder Cancer (NMIBC)
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor's decision
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Collaborators: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A9EO9201; EO9_C301
Record Dates: First submitted 2011-11-16; First posted 2011-11-21 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2013-04

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; NMIBC; TURBT; Apaziquone; EOquin; Immediate instillation
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — apaziquone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EO9 (Apaziquone) (Experimental)
  Interventions: Drug: EO9 (Apaziquone)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EO9 (Apaziquone) — 4 mg/40 mL, Intravesical instillation, Single dose within 6 hours after TURBT
  Other Names: Eoquin(R)
  Arms: EO9 (Apaziquone)
Drug: Placebo — 40 mL, Intravesical instillation, Single dose within 6 hours after TURBT
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety in patients with non-muscle invasive bladder cancer histologically diagnosed to be stage Ta and G1 or G2 and who were randomized into either an EO9 or placebo group after TURBT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have provided written informed consent
2. Patients who have urothelial cell carcinoma of the bladder with clinically apparent stage Ta, grade G1-G2 and satisfy both of the following criteria:

   * The maximum number of tumors is 5.
   * Each tumor diameter: ≤ 3.5 cm.
3. Age: ≥20 years old at enrollment.
4. The functions of the major organs are adequate, and the following test value criteria are satisfied:

   * Neutrophil count ≥1,500/μL
   * Platelet count ≥10×10^4/μL
   * Hemoglobin ≥10 g/dL

Exclusion Criteria:

1. Patients with a single, primary bladder cancer of <0.5 cm.
2. Patients with CIS lesions in the bladder or a history thereof.
3. Patients with a history of other than stage Ta, histological grade G1 or G2 disease.
4. Patients experiencing recurrence within 4 months following TURBT for prior NMIBC (duration between the last TURBT and cystoscopic confirmation of the present recurrence is within 4 months).
5. Patients without at least a three-month cystoscopically confirmed recurrence-free interval between the last TURBT and the time of study screening
6. Patients having a bladder tumor with a histological diagnosis other than urothelial carcinoma of the bladder or a history thereof.
7. Patients who had been administered EO9 in the past.
8. Patients who had been administered any other investigational drug within the past 30 days.
9. Patients having a medical condition that would make it unsafe for them to undergo TURBT under general or spinal anesthesia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
The recurrence rate at 2 years in patients with histologically diagnosed stage Ta, grade G1 or G2 bladder cancer | 2 years

SECONDARY OUTCOMES:
The recurrence-free interval in patients with histologically diagnosed stage Ta, grade G1 or G2 bladder cancer | 2 years
The progression rate | 2 years
The number of recurrences per patient | 2 years
The progression-free survival period | 2 years
The recurrence-free survival period | 2 years
The overall survival period | 2 years
The safety of EO9 | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yoshihiro Nambu, M.D., Ph.D., Study Director — Nippon Kayaku Co., Ltd.; Woo Ick Jang, M.D., Ph.D., Study Director — Handok Inc.
Locations (20):
- Japan (11):
  - Nippon Kayaku Investigational site 103, Yokosuka, Kanagawa
  - Nippon Kayaku Investigational site 107, Kashihara, Nara
  - Nippon Kayaku Investigational site 109, Kurashiki, Okayama-ken
  - Nippon Kayaku Investigational site 105, Sayama, Osaka
  - Nippon Kayaku Investigational site 104, Hamamatsu, Shizuoka
  - Nippon Kayaku Investigational site 102, Musashino, Tokyo
  - Nippon kayaku Investigational site 101, Chiba
  - Nippon Kayaku Investigational site 110, Fukuoka
  - Nippon Kayaku Investigational site 111, Fukuoka
  - Nippon Kayaku Investigational site 106, Nara
  - Nippon Kayaku Investigational site 108, Okayama
- South Korea (9):
  - Handok Investigational site 203, Bundang
  - Handok Investigational site 202, Daegu
  - Handok Investigational site 209, Hwasun
  - Handok Investigational site 201, Seoul
  - Handok Investigational site 204, Seoul
  - Handok Investigational site 205, Seoul
  - Handok Investigational site 206, Seoul
  - Handok Investigational site 207, Seoul
  - Handok Investigational site 208, Yangsan